CLINICAL TRIAL: NCT05955690
Title: Knowledge and Attitude of Pregnant Women Towards Preeclampsia and Its Associated Factors in Assuit University Women's Health Hospital.
Brief Title: Knowledge and Attitude of Pregnant Women Towards Preeclampsia in Assiut Governorate
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Khalaf Refaey, Principle investigator, Assiut University
Other Study IDs: gehadkhalaf
Record Dates: First submitted 2023-07-12; First posted 2023-07-21 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2024-09

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Our study will be a cross sectional study to evaluate the knowledge level and attitude of pregnant women towards preeclampsia and factors affecting it ,the study will be done at Assiut University Hospitals - Women's Health Hospital. all pregnant women who will come to ANC visits will be included .the study tool is a well structured questionnaire for assessment of our outcomes.

DETAILED DESCRIPTION:
Preeclampsia is a pregnancy-related hypertensive disorder that usually occurs after 20 weeks of gestation. It is characterised by hypertension and proteinuria . Preeclampsia is the leading cause of maternal death, complicating about one-tenth of all pregnancies worldwide . It is the second greatest cause of direct maternal death, accounting for 70,000 maternal mortality globally each year .The burden of preeclampsia and eclampsia is most significant in low- and middle-income countries (LMICs), where hypertensive disorders of pregnancy account for 10-15% of maternal deaths.

Early detection of symptoms, rapid presentation to healthcare facilities, and subsequent management with antihypertensive medications, magnesium sulphate, and delivery of the foetus and placenta improve outcomes in pregnancies complicated by preeclampsia and eclampsia . As a result, ANC visits and intrapartum admission are critical chances for patient counselling Despite the essential relationship between women's awareness of preeclampsia and health seeking behaviour, research on this topic is limited, particularly in underdeveloped countries. Even in developed countries, studies in high-income countries show that only half of patients were counselled about preeclampsia signs and symptoms, despite the fact that counselling by healthcare personnel is related to higher patient knowledge. So there is a gap in studying pregnant women's knowledge and attitudes concerning preeclampsia in underdeveloped countries, particularly Egypt, where studies on this topic are scarce.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women.
* pregnant women in first, second and third trimester.
* pregnant women who come to receive ANC at Assiut University Hospitals - Women's Health Hospital out patient clinic.

Exclusion Criteria:

* Pregnant women that are unwell to give consent.
* Pregnant women who are already diagnosed by preeclampsia and eclampsia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — because we need pregnant women so it is a gender based study
Study Population: All pregnant women in first, second and third trimester who will come to receive antenatal care (ANC) services
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Knowledge of pregnant women about preeclampsia | just after ending the interview in which we filled in questionnaire
  assessement of knowledge"poor,moderate or good " by answering a structured questionnaire .The women will answer by yes , no or I don't know , A scoring system, where a correct answer attracts a score of one (1) and a wrong or no response (or I don't know) attracts a score of zero (0) was used to scale participants' knowledge of preeclampsia . The scores were expressed as percentages and Bloom's cut-off point will be employed to classify knowledge of PE into three levels: poor (< 60%), moderate (60-80%) and good (80-100%).high score means a better outcome .
Attitude of pregnant women towards preeclampsia | just t after ending the interview in which we filled in questionnaire
  assessement of attitude ""positive ,neutral or negative " by answering a structured questionnaire.The women will answer by agree ,disagree or unsure , Attitude was reported as positive, neutral and negative when they scored 80-100 %, 60-79 %, and less than 60 % of the attitude assessment questions respectively using the Bloom's cut-off point.
Associated factor with knowledge and attitude of pregnant women towards preeclampsia | through study completion, an average of 1 year
  studying sociodemographic ,medical and obstetric factors that affect knowledge and attitude of pregnant women towards preeclampsia by well structured questionnaire "by the previous scale"

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abbas, MD, Study Chair — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No